CLINICAL TRIAL: NCT04070807
Title: Italian Observational Study of Patients With Acute Myeloid Leukemia Treated With Small Molecule Inhibiting B-cell Lymphoma 2 (BCL-2)
Brief Title: Italian Observational Study of Patients With Acute Myeloid Leukemia Treated With Small Molecule Inhibiting BCL-2
Acronym: AVALON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IRST204.04
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; BCL-2; anti BCL2 inhibitors; clinical practice
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center retrospective observational study. Every patient with Acute Myeloid Leukemia (AML) treated with anti-B-cell lymphoma 2 (BCL2) treatment outside clinical trial from 1st January 2015 up to 01 April 2019 may be included in this study. No additional drug/procedures/patient visits in comparison with the usual clinical practice are planned for the study. The decision to treat patient with ant-BCL2 inhibitors is made by the physician based on his clinical judgment, independently from the decision to include the patient in this study.

DETAILED DESCRIPTION:
In phase 1-2 studies, anti BCL-2 treatment has shown evidence of anti-leukemic activity as single agent and in combination and proved to be particularly effective in providing a deep response, with an acceptable safety profile. Since 2015 anti-BCL2 treatment has been available in other indications and in off-label use in Italy.

In this non-interventional retrospective study, toxicity, effectiveness and costs assessment data will be collected from patients with AML, to improve the knowledge about anti-BCL2 treatment in clinical practice. Collecting and analyzing data from a large unbiased patient-set receiving anti-BCL2, would enlarge our knowledge on therapies inhibiting BCL2.

This is a multi-center retrospective observational study. Every patient with AML treated with anti-BCL2 treatment outside clinical trial from 1st January 2015 up to 01 April 2019 may be included in this study. No additional drug/procedures/patient visits in comparison with the usual clinical practice are planned for the study. The decision to treat patient with ant-BCL2 inhibitors is made by the physician based on his clinical judgment, independently from the decision to include the patient in this study. As this study is intended to be purely observational (not interventional), the patient's medical records will be the source of all data to be recorded. No additional procedures/patient visits should be planned in the study with respect to clinical practice.

Clinical data (treatment, survival, adverse events) will be collected for patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patient with AML according to World Health Organization (WHO) 2016 classification
* Patient who have received any anti-BCL-2 treatment as single agent or in combination with other drugs from 1 Jan 2015 to 1 Apr 2019 outside clinical trials

Exclusion Criteria:

• Patient who have received any anti-BCL-2 treatment within a clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AML according to World Health Organization (WHO) 2016 classification who have received any anti-BCL-2 treatment as single agent or in combination with other drugs from 1 Jan 2015 to 1 Apr 2019 outside clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events of grade 3 and 4 (NCTCAE version 5.0) | up to 18 months
  To evaluate the toxicity profile of the therapy with anti-BCL-2 in patients with AML.

SECONDARY OUTCOMES:
Overall Survival | 18 months
  to describe the clinical outcomes in terms of Overall Survival (OS) defined as the number of days between the first study drug administration and death from any cause
Disease Free Survival (DFS) | 18 months
  to describe Disease Free Survival, defined as the number of days between the first study drug administration and any event including disease progression or death from any cause (both median and restricted mean) whichever occurs first.
Complete Remission | 18 months
  to describe the Complete Remission (CR), in terms of proportions, in response to therapy
Complete Remission with incomplete hematologic recovery | 18 months
  to describe Complete Remission with incomplete hematologic recovery (CRi) in terms of proportions, in response to therapy
Minimal Residual Disease | 18 months
  to describe Minimal Residual Disease, in terms of proportions, in response to therapy
Incidence of successful bridge to allogeneic transplant | 18 months
  to describe the incidence of successful bridge to allogeneic transplant, in terms of proportions, in response to therapy
Collection of number of hospitalizations | 18 months
  to describe healthcare resource utilization in terms of number of hospitalizations per patient
Collection of days of hospitalizations | 18 months
  to describe healthcare resource utilization in terms of days of hospitalizations per patient
Collection of number of clinical visits per patient | 18 months
  to describe healthcare resource utilization in terms of number of clinical visits per patient
Collection of number of accesses Day Hospital per patient | 18 months
  to describe healthcare resource utilization in terms of number of accesses in Day Hospital per patient
Collection of number of accesses in Emergency Care Units per patient | 18 months
  to describe healthcare resource utilization in terms of number of accesses in Emergency Care Units per patient

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Principal Investigator — IRST IRCCS
Locations (20):
- Italy (20):
  - ASST Cremona, Cremona, CR
  - A.O. Pugliese Ciaccio, Catanzaro, CZ
  - Irst Irccs, Meldola, FC
  - AOU Careggi, Florence, FI
  - IRCCS Casa Sollievo sofferenza, San Giovanni Rotondo, Foggia
  - Ospedale F. Spaziani, Frosinone, FR
  - P.O. Vito Fazzi, Lecce, LE
  - Ospedale Santa Maria Goretti, Latina, LT
  - Asst Monza, Monza, MB
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Ospedale S.Spirito - ASL Pescara, Pescara, PE
  - Ospedale Santa Maria della Misericordia, Perugia, PG
  - AOU San Giovanni di Dio e Ruggi D'Aragona, Salerno, SA
  - Policlinico Santa Maria alle Scotte, Siena, SI
  - AOU Città della Salute e della Scienza di Torino, Torino, TO
  - A.O. Ordine Mauriziano, Torino, TO
  - Ospedale Ca' Foncello, Treviso, TV
  - European Institute of Oncology, Milan
  - Fondazione IRCCS Ca' Granda OSPEDALE MAGGIORE POLICLINICO, Milan
  - Ospedale Roma S.Eugenio, Roma

IPD SHARING:
Plan to Share IPD: No